CLINICAL TRIAL: NCT02632253
Title: Effects of High-intensity Interval Training on Exercise Capacity in Patients With Grown-up Congenital Heart Disease (GUCH)
Brief Title: Effects of High-intensity Interval Training on Exercise Capacity in Patients With Grown-up Congenital Heart Disease
Acronym: HIIT-GUCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patients recruited due to a lack of GUCH patients enrolling in cardiac Rehabilitation.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Schweizerische Herzstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT-GUCH
Record Dates: First submitted 2015-12-02; First posted 2015-12-16 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Congenital Heart Defects
Keywords: exercise therapy; GUCH; ventricular ejection fraction; HIIT; MICE
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate intensity continuous exercise (Active Comparator): Patients perform two weekly supervised MICE session on a cycling ergometer per week plus one self monitored 30-60 min MICE training of choice at home.
  MICE is performed on a cycle ergometer at an intensity of 70-75% of peak heart rate for 38 min (including a 5 min warm-up and 3 min cool-down).
  Interventions: Other: MICE
- High intensity interval training (Experimental): High-intensity interval training (HIIT) is performed on a cycle ergometer. It consists of a 10 min warm-up followed by 4 min intervals in Zone III (at 90-95% of peak heart rate), with each interval separated by 3 min of active pauses in zone I (at 50-70% of peak heart rate). The total duration of the HIIT training is 38 min.
  Additionally patients perform one self monitored 30-60 min MICE training of choice per week at home.
  Interventions: Procedure: HIIT

INTERVENTIONS:
Procedure: HIIT — High-intensity interval training (HIIT) is performed on a cycle ergometer. It consists of a 10 min warm-up followed by 4 min intervals in Zone III (at 90-95% of peak heart rate), with each interval separated by 3 min of active pauses in zone I (at 50-70% of peak heart rate). The total duration of the HIIT training is 38 min. The HIIT group will perform two supervised HIIT trainings and one self monitored MICE training per week.
  Arms: High intensity interval training
Other: MICE — MICE is also performed on a cycle ergometer at an intensity of 70-75% of peak heart rate for 47 min (in order for the two training protocols to be isocaloric). The control group will perform two supervised and one self monitored MICE training per week.
  Arms: Moderate intensity continuous exercise

SUMMARY:
Patients with congenital heart disease have long been discouraged from participating in physical exercise which has led to impaired exercise capacity in this population. Since low physical and cardiorespiratory fitness has been shown to be a predictor for hospitalization and mortality in grown-up patients with congenital heart disease (GUCH), aerobic endurance training has been recommended recently to improve exercise capacity. The aim of this study is to compare two types of training, namely high-intensity interval training (HIIT) and moderate-intensity continuous exercise (MICE), with regard to improving exercise capacity without adverse effects on heart structure, function and rhythm in the setting of a 12-week outpatient cardiac rehabilitation (CR) program in GUCH with a remaining pathology involving the right and/or left ventricles. Primary endpoint will be change in exercise capacity (maximal oxygen consumption) over the 12-week CR. Secondary endpoints will be changes of the right or left ventricles as well as vascular function.

Patients with GUCH and reduced function of the right ventricle will be recruited and informed about the study within the first two weeks of CR. At the end of week 3 of the CR with supervised MICE, randomization to 9 weeks of twice weekly either HIIT or MICE takes place.

MICE training is performed at an intensity of 70-85% of maximum heart rate (HRmax) for 38 min. HIIT consists of four 4 min bouts of high-intensity exercise (90-95% of HRmax), interspersed by 3 min low-intensity intervals (50-60% of HRmax). All patients complete one additional endurance activity per week in their own time with a duration of 30-60 min at moderate intensity monitored by their smart phone.

Change in peak oxygen uptake as well as maximal exercise capacity at the end of an incremental cardiopulmonary exercise test will be assessed between week 3 and 12. Vascular function will be assessed at the same time. Volumes and function of the right and left ventricles will be measured by cardiac magnetic resonance imaging (CMR) upon inclusion into the study and at completion of the intervention. Furthermore, laboratory markers for heart failure as well as occurrence of irregular fast heart beats will be assessed.

DETAILED DESCRIPTION:
Background

Adults with congenital heart disease have long been recommended to refrain from physical exercise. Therefore, they often have significant reduction in exercise capacity. Only recently, regular exercise has been shown to be safe and is nowadays recommended for patients with congenital heart disease. As a result, exercise based rehabilitation programs have been implemented in order to improve exercise capacity and avoid adverse effects associated with inactive lifestyle.

Several studies have shown that high-intensity interval training (HIIT) is more effective than moderate-intensity continuous exercise training (MICE) at improving functional capacity and quality of life in stable cardiac patients and can be performed safely. It has therefore emerged as a new and important exercise modality in cardiac rehabilitation centers all over Europe for stable cardiac patients with left ventricular (LV) dysfunction. However, its safety and efficacy has not yet been tested in adults with congenital heart disease and to date there are no studies who have evaluated whether short term peaks of pulmonary artery or systemic pressure during bouts of 4 min of high-intensity exercise negatively affects the subpulmonary or systemic ventricle in GUCH patients. The investigators hypothesized that the positive effects of HIIT on exercise capacity and vascular function found in patients with ischemic cardiomyopathy can be transferred to the population of GUCH patients, and that short-term bouts of high-intensity exercise will not negatively affect cardiac morphology and function.

Objective

To test the superiority of a 9-week high-intensity interval training (HIIT) over a standard rehabilitation training based on moderate-intensity continuous exercise (MICE) on exercise capacity in patients with grown-up congenital heart disease (GUCH) with a residual pathology involving the right and/or left ventricle (RV/LV).

Methods

Measurements will be performed before and after a 12 week intervention with either HIIT or MICE training. Patients will undergo cardiopulmonary exercise testing on a cycle ergometer to determine exercise capacity and VO2 peak. Cardiac magnetic resonance imaging will be performed for ventricular volumes, mass and function. Vascular function will be assessed by arterial stiffness measurement. Physical exercise, quality of life will be evaluated by questionnaires.

During the 4th and the 12th week of the rehabilitation training, heart rate variability will be measured in the morning following a training, and blood samples will be taken after a training session to analyse markers of myocardial stress (hs Troponin and N-terminal of the prohormone brain natriuretic peptide, NT pro-BNP). Compliance and acceptance of training will be assessed by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Tetralogy of Fallot
* Double outlet right ventricle
* Transposition of the great arteries with atrial or arterial switch
* Treated or untreated pulmonary valvular or pulmonary artery stenosis
* Reduced right ventricular function after correction of atrial septal defect (ASD), atrio-ventricular septal defect (AVSD) or ventricular septal defect (VSD) (≤40%)
* Ebstein anomaly
* Patients with a systemic right ventricle like d-transposition of the great arteries (d-TGA) with previous atrial switch operation or cc-TGA

Exclusion Criteria

* Inability to participate in a 3-month training program in Bern
* New York Heart Association class ≥ III
* Ventricular function ≤30% of either the systemic or the sub-pulmonary ventricle
* Moderate to severe LV outflow tract obstruction (valvular, subvalvular, due to asymmetric septum hypertrophy, or aortic coarctation) with mean gradient >30 mmHg by echo
* Severe RV outflow tract obstruction with peak gradient ≥60 mmHg by echo
* Moderate to severe pulmonary hypertension with mean pulmonary artery pressure≥40 mmHg
* Resting saturation at ambient air of <90%
* Pacemaker or Implantable Cardioverter Defibrillator
* Contraindication to perform a CMR (cerebral clips, iron-containing body implants, medical pumps)
* Recent episode of ventricular tachycardia
* Permanent atrial fibrillation
* Unstable angina or recent myocardial infarction (<12 months)
* Recent cardiac operation <6 months
* Ascending aortic dilatation >45 mm in patients with bicuspid aortic valve or >50 mm in patients without bicuspid aortic valve
* Repaired coarctation with pseudoaneurysm in MR angiography
* No consent
* Any medical condition which would prevent a patient from performing high intensity training (e.g. cardiac thrombus formation, recent valve surgery (< 1 year), in general orthopedic, peripheral vascular, neurologic or other limitations)
* Inability to perform cardiopulmonary exercise testing
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2 peak) during maximal cardiopulmonary exercise test | week 1 to 12
  Change in VO2 peak between week 1 and 12 is measured by cardiopulmonary exercise testing on a cycling ergometer.

SECONDARY OUTCOMES:
VO2 peak during maximal cardiopulmonary exercise test | week 1 to 65
  Change in VO2 peak between week 1 and 65 is measured by cardiopulmonary exercise testing on a cycling ergometer.
Ventricular Volumes by cardiac magnetic resonance imaging | week 1 and 12
  Left and right ventricular volumes will be assessed by cardiac magnetic resonance imaging.
Ventricular function by cardiac magnetic resonance imaging (MR) | week 1 and 12
  Left and right ventricular function will be assessed by cardiac magnetic resonance imaging (MR).
Vascular function by arterial stiffness measurement | week 3, 12, and 65
  Vascular function will be assessed by arterial stiffness measurement.
Arrhythmias quantified and characterised by ECG | week 3, 12, and 65
  Arrhythmias will be assessed by 24-hour Holter ECG.
N terminal pro b-type natriuretic peptide (NT- proBNP) | week 0, 3, 12, and 65
  Blood samples are taken after an exercise training session.
hs Troponin | week 3 and 12
  Blood samples are taken after an exercise training session.
Adherence to training | week 1-12
  Training session adherence will be monitored and reported as percent of prescribed training volume.
Quality of life | week 1, 12, and 65
  Short form quality of life questionnaire (SF12)
Quality of life for heart failure | week 1, 12, and 65
  Minnesota quality of life questionnaire
Daily physical activity | week 1, 12, and 65
  International physical activity questionnaire
Heart rate variability | week 3, 12, and 65
  Heart rate variability will be assessed during an orthostatic challenge test.

OTHER OUTCOMES:
Heart rate variability | week 3 and 12
  Heart rate variability will be measured overnight and in the morning after a day with a training session and after a day without training.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Deluigi, MD, Principal Investigator — Preventive Cardiology & Sports Medicine, University Clinic for Cardiology, University Hospital Berne, Inselspital, Bern, Switzerland
Locations (1):
- Department of Preventive Cardiology, Bern University Hospital, Bern, Switzerland